CLINICAL TRIAL: NCT05958121
Title: A Phase I/II First-In-Human Clinical Trial to Evaluate the Safety, Tolerability and Anti-Tumor Activity of IMA402, a Bispecific TCER® Targeting PRAME, in Patients With Recurrent and/or Refractory Solid Tumors
Brief Title: IMA402 T Cell-Engaging Receptor Molecule (TCER®) in Recurrent and/or Refractory Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immatics Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMA402-101; 2022-503133-54-00 (Other: Clinical Trials Information System)
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Refractory Cancer; Recurrent Cancer; Solid Tumor, Adult; Cancer
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation/de-escalation (Phase Ia) (Experimental): Dose-Finding of IMA402 (Phase Ia)
  Interventions: Biological: IMA402 (Phase Ia)
- Dose extension (Phase Ib) (Experimental): IMA402 monotherapy extension cohorts based on maximum tolerated dose (MTD) and/or recommended doses for extensions (RDEs) (Phase Ib)
  Interventions: Biological: IMA402 (Phase Ib)
- Dose extension (Phase II) (Experimental): Selected ISEC investigated on MTD/RDEs based on a manageable/favorable safety profile and initial signs of anti-tumor activity (Phase II)
  Interventions: Biological: IMA402 (Phase II)

INTERVENTIONS:
Biological: IMA402 (Phase Ia) — Intravenous infusions in escalating dose levels
  Arms: Dose escalation/de-escalation (Phase Ia)
Biological: IMA402 (Phase Ib) — Treatment at MTD and/or RDE (Phase Ib)
  Arms: Dose extension (Phase Ib)
Biological: IMA402 (Phase II) — Treatment at MTD/RDE based on a manageable/favorable safety profile and initial signs of anti-tumor activity of selected ISEC (Phase II)
  Arms: Dose extension (Phase II)

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and anti-tumor activity of IMA402 in patients with recurrent and/or refractory solid tumors.

Primary objectives:

* To determine the maximum tolerated dose and/or recommended dose for extension for IMA402 (Phase I)
* To characterize the safety and tolerability of IMA402 (Phase I/II)
* To evaluate anti-tumor activity of IMA402 (Phase II)

Secondary objectives:

* To evaluate the initial anti-tumor activity of IMA402 (Phase I)
* To evaluate anti-tumor activity of IMA402 (Phase II)
* To describe the PK of IMA402 (Phase I/II)

DETAILED DESCRIPTION:
The study will be conducted in two phases:

* Phase Ia: Dose escalation/de-escalation
* Phase Ib: Dose extension
* Phase II: Dose extension in selected Indication-specific extension cohort(s) (ISEC)

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients must have a specific pathologically confirmed and documented advanced and/or metastatic solid tumor indication
* Patients must have received or not be eligible for all available indicated standard-of-care treatments
* Measurable disease according to RECIST 1.1
* Confirmed HLA status
* ECOG Performance Status of 0 to 1
* Adequate baseline hematologic, hepatic and renal function, acceptable coagulation status

Exclusion Criteria:

* Other active malignancies that require treatment or that might interfere with the trial endpoints (ongoing adjuvant anti-hormonal treatment is allowed)
* The patient is pregnant or is breastfeeding
* History of hypersensitivity to components of IMA402 or rescue medications, if no alternative treatment option is available
* The patient has concurrent severe and/or uncontrolled medical disease. Any other health condition that would, in the investigator's judgement, contraindicate the patient's participation in the clinical trial because of safety concerns or compliance with clinical trial procedures
* Patients with active brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Phase I: Number of patients with dose limiting toxicities (DLTs) | 24 months
Phase I/II: Number of patients with treatment-emergent adverse events (TEAEs) | 40 months
Phase I/II: Number of patients with serious TEAEs | 40 months
Phase I/II: Frequency of dose interruptions and reductions, permanent discontinuations | 40 months
Phase I/II: Duration of dose interruptions and reductions, permanent discontinuations | 40 months
Phase II: Overall response rate (ORR) based on best overall response (BOR) of complete response (CR) and partial response (PR) locally assessed using Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) | 40 months

SECONDARY OUTCOMES:
Phase I: ORR based on BOR of CR and PR locally assessed using RECIST v1.1 and iRECIST | 37 months
Phase II: ORR based on BOR of CR and PR locally assessed using iRECIST | 40 months
Phase I/II: Disease control rate (DCR) of CR, PR or stable disease (SD) (lasting 6 or more weeks) following the initiation of IMA402 based on RECIST v1.1 and iRECIST | 40 months
Phase I/II: Duration of response (DOR) of CR or PR based on RECIST v1.1 and iRECIST | 40 months
Phase I/II: Progression-free survival (PFS) based on RECIST v1.1 and iRECIST | 40 months
Phase I/II: Overall survival (OS) | 40 months
Phase I/II: Determination of PK parameter: half-life (t1/2) | 40 months
Phase I/II: Determination of PK parameter: minimal serum concentration (Cmin) | 40 months
Phase I/II: Determination of PK parameter: maximal serum concentration (Cmax) | 40 months
Phase I/II: Determination of PK parameter: area under the curve (AUC) | 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Immatics Biotechnologies GmbH, Study Director — Immatics Biotechnologies GmbH
Locations (24):
- Germany (20):
  - Universitaetsklinikum Heidelberg AöR, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm AöR, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen AöR, Erlangen, Bavaria
  - Klinikum Nürnberg, Nuremberg, Bavaria
  - Universitaetsklinikum Regensburg, Regensburg, Bavaria
  - Universitaetsklinikum Wuerzburg AöR, Würzburg, Bavaria
  - Justus-Liebig-Universitaet Giessen, Giessen, Hesse
  - Philipps-Universitaet Marburg, Marburg, Hesse
  - Elbe Kliniken Stade- Buxtehude Elbe Klinikum Buxtehude gGmbH, Buxtehude, Lower Saxony
  - Universitaetsklinikum Bonn AöR, Bonn, North Rhine-Westphalia
  - Marien Hospital Duesseldorf GmbH, Düsseldorf, North Rhine-Westphalia
  - KEM I Evang. Kliniken Essen-Mitte gGmbH, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Essen AöR, Essen, North Rhine-Westphalia
  - Johannes Wesling Klinikum Minden, Minden, North Rhine-Westphalia
  - Universitaet Muenster, Münster, North Rhine-Westphalia
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universitaetsklinikum Carl Gustav Carus Dresden an der Technischen Universitaet Dresden AöR, Dresden, Saxony
  - University Of Leipzig, Leipzig, Saxony
  - Universitaetsklinikum Magdeburg AöR, Magdeburg, Saxony-Anhalt
- Netherlands (4):
  - Antoni von Leeuwenhoek- Netherlands Cancer Institute, Amsterdam, North Holland
  - Leiden Universitair Medisch Centrum, Leiden, South Holland
  - Universitair Medisch Centrum Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- See also: Corporate Website — http://immatics.com/